CLINICAL TRIAL: NCT05242952
Title: LEveraging A viRtual eNvironment (LEARN) to Enhance Prevention of HIV-related Comorbidities in At-risk Minority MSM
Brief Title: The LEARN Study for CVD Prevention
Acronym: LEARN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000031403; 1K01HL145580-01A1 (NIH)
Record Dates: First submitted 2020-10-28; First posted 2022-02-16 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Cardiovascular Diseases
Keywords: Comorbidity; Cardiovascular Diseases; Sexual and Gender Minorities; HIV Infections; Virtual Reality; Cardiovascular Health
MeSH Terms: conditions — Cardiovascular Diseases; Coitus; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention Group (Experimental): Participants will enter an online game and learn about how to prevent cardiovascular and metabolic conditions.
  Interventions: Behavioral: Gaming in a virtual environment
- Waitlist Control Group (Other): Participants will enter an online game at a later date after the immediate intervention group and learn about how to prevent cardiovascular and metabolic conditions.
  Interventions: Behavioral: Gaming in a virtual environment

INTERVENTIONS:
Behavioral: Gaming in a virtual environment — To address the primary outcomes of feasibility and acceptability of the VE, we will capture process data using a computer-based virtual environment and self-report measures using an online survey.

SUMMARY:
The investigator is testing a virtual environment to address prevention of HIV-related comorbidities.

DETAILED DESCRIPTION:
The primary aims of this study are to test the feasibility, acceptability and preliminary effects of a VE to address prevention of HIV-related comorbidities. A waitlist control feasibility clinical trial will be conducted. We will assign (N=80) eligible participants and ensure balanced allocation to intervention and control groups over the intervention period. We hypothesize that the VE will be feasible and acceptable to persons living with HIV, and that they will apply their VE learning to real-life situations and health behaviors for prevention of HIV-related comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* identify as an ethnic/racial minority with HIV
* identify as gay, same-gender-loving, or MSM
* able to read and understand English
* access to a computer capable of downloading and running the VE software
* no medical history of serious cardiovascular or cognitive complications

Exclusion Criteria:

Anything outside of inclusion parameters, including history of:

* myocardial infarction (MI)
* congestive heart failure (CHF)
* coronary artery bypass graft (CABG)
* cerebral vascular accident (CVA)
* cognitive impairment

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — assigned male sex at birth
Enrollment: 78 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Acceptability/Feasibility {change over 3 timepoints} | Baseline and Month 3 & 6
  Based on Technology Acceptance Model, using the same unit of measure, we will examine Perceived Usefulness (Cronbach's alpha 0.98) and Perceived Ease of Use (Cronbach's alpha 0.94) with an online 7-point Likert scale.

SECONDARY OUTCOMES:
Cardiovascular health {change over 3 timepoints} | Baseline and Month 3 & 6
  Life's Simple 7, based on 7 modifiable health behaviors, provides scores (range, 0 to 14) based on smoking, diet, physical activity, body mass index, blood pressure, total cholesterol, and fasting glucose. This study will only measure 4 out of the 7: smoking, diet, physical activity, and BMI.
Physical Activity {change over 3 timepoints} | Baseline and Month 3 & 6
  International Physical Activity Questionnaire - Short Form will assess intensity of physical activity and sitting time using a 7-item, open-ended measure. Cronbach's alpha 0.80.
Tobacco and E-cigarette use {change over 3 timepoints} | Baseline and Month 3 & 6
  BRFSS - self report measure questions that pertain to Tobacco use and E-cigarette use (7 questions). kappa statistic 0.81-0.92.
Food consumption {change over 3 timepoints} | Baseline and Month 3 & 6
  Food Frequency Questionnaire - Reports how frequently individuals consume foods in 16 categories. Multifactor Screener has demonstrated correlations of 0.5-0.8 with estimated true intake.
Psychosocial wellbeing {change over 3 timepoints} | Baseline and Month 3 & 6
  Patient Health Questionnaire-9. PHQ-9 is a 9-item validated questionnaire used to screen for depression with a range of scores from 0-45. A cumulative score of ≥10 is considered positive with lower scores indicating no or mild anxiety.
Illness Perceptions {change over 3 timepoints} | Baseline and Month 3 & 6
  The Revised Illness Perception Questionnaire measures illness perceptions about hypertension and type 2 diabetes on a 5-point Likert scale ("strongly disagree" to "strongly agree").

CONTACTS AND LOCATIONS:
Overall Officials: S. Raquel Ramos, PhD, MBA, MSN, FNP-BC, Principal Investigator — Yale University School of Nursing
Locations (1):
- Yale University, Orange, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramos SR, Warren R, Shedlin M, Melkus G, Kershaw T, Vorderstrasse A. A Framework for Using eHealth Interventions to Overcome Medical Mistrust Among Sexual Minority Men of Color Living with Chronic Conditions. Behav Med. 2019 Apr-Jun;45(2):166-176. doi: 10.1080/08964289.2019.1570074. PMID 31343963
- [Background] Ramos SR, O'Hare OM, Hernandez Colon A, Kaplan Jacobs S, Campbell B, Kershaw T, Vorderstrasse A, Reynolds HR. Purely Behavioral: A Scoping Review of Nonpharmacological Behavioral and Lifestyle Interventions to Prevent Cardiovascular Disease in Persons Living With HIV. J Assoc Nurses AIDS Care. 2021 Sep-Oct 01;32(5):536-547. doi: 10.1097/JNC.0000000000000230. PMID 33481464
- [Background] Ramos SR, Johnson C, Melkus G, Kershaw T, Gwadz M, Reynolds H, Vorderstrasse A. Cardiovascular Disease Prevention Education Using a Virtual Environment in Sexual-Minority Men of Color With HIV: Protocol for a Sequential, Mixed Method, Waitlist Randomized Controlled Trial. JMIR Res Protoc. 2022 May 17;11(5):e38348. doi: 10.2196/38348. PMID 35579928
- [Result] Ramos SR, Reynolds H, Johnson C, Melkus G, Kershaw T, Thayer JF, Vorderstrasse A. Perceptions of HIV-Related Comorbidities and Usability of a Virtual Environment for Cardiovascular Disease Prevention Education in Sexual Minority Men With HIV: Formative Phases of a Pilot Randomized Controlled Trial. J Med Internet Res. 2024 Aug 22;26:e57351. doi: 10.2196/57351. PMID 38924481